CLINICAL TRIAL: NCT02842021
Title: A Randomized, Double-Blind, Active- and Vehicle-Controlled Study to Compare the Efficacy and Safety of Products S2G6T-1, S2G6T-2, S2G6T-3 and S2G6T-4 in Patients With Symptomatic Inflammatory Interdigital Tinea Pedis
Brief Title: Efficacy and Safety of Product S2G6T-1in Patients With Symptomatic Inflammatory Interdigital Tinea Pedis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Failed to meet success criteria
Sponsor: Sol-Gel Technologies, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SGT-26-01
Record Dates: First submitted 2016-07-13; First posted 2016-07-22 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Tinea Pedis
MeSH Terms: conditions — Tinea Pedis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- S2G6T-1 (Active Comparator): Topical cream
  Interventions: Drug: S2G6T-1
- S2G6T-2 (Active Comparator): Topical Cream
  Interventions: Drug: S2G6T-2
- S2G6T-3 (Active Comparator): Topical Cream
  Interventions: Drug: S2G6T-3
- S2G6T-4 (Placebo Comparator): Topical Cream
  Interventions: Drug: S2G6T-4

INTERVENTIONS:
Drug: S2G6T-1 — Twice a day topical cream
  Arms: S2G6T-1
Drug: S2G6T-2 — Twice a day topical cream
  Arms: S2G6T-2
Drug: S2G6T-3 — Twice a day topical cream
  Arms: S2G6T-3
Drug: S2G6T-4 — Twice a day topical cream
  Arms: S2G6T-4

SUMMARY:
To assess the efficacy and safety of a combination product S2G6T-1 compared to its monads and vehicle, applied twice daily for 7 days, in the treatment of symptomatic inflammatory interdigital tinea pedis in subjects 12 years of age and older. The results of this study will be utilized to perform power calculations for the Phase 3 pivotal trials.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to sign a written informed consent and /or assent (age appropriate).
2. Male or Female subjects 12 years of age or older.
3. A clinical diagnosis of interdigital tinea pedis on one or both feet characterized by clinical evidence of a tinea infection.
4. A sum of at least five (5) for signs (erythema and scaling) by the investigator on the selected target foot, and a score of at least five (5) for each symptom: pruritus (itching) and burning: and a sum of at least twelve (12) for both symptoms (pruritus and burning) by the subject on the PATSS.
5. Mycological evidence of the presence of fungi confirmed by the detection of fungal hyphae on a microscopic KOH wet mount.
6. Females of child-bearing potential must have a negative urine pregnancy test and must agree to use an effective form of contraception during the study .
7. Must be in good general health as determined by medical history and free of any disease that in the investigator's opinion might interfere with the study evaluations.
8. Must be able to communicate, be able to understand the study procedures, and be willing to comply with the study requirements.

Exclusion Criteria:

1. The presence of confluent diffuse moccasin-type tinea pedis.
2. Negative KOH microscopy test to assess presence of hyphae.
3. Onychomycosis of the toenails, involving ≥ 20% of the area of either great toenail or involvement of more than five toenails in total.
4. Concurrent tinea infection or bacterial skin infection on the feet.
5. Female subjects who are pregnant and/or nursing or planning a pregnancy during the course of the trial.
6. Recent history of or currently known to abuse drugs or alcohol.
7. History of intolerance or hypersensitivity to Econazole Nitrate, Mometasone Furoate, or other imidazole agents.
8. Presence of any other infection of the foot or other disease process that might confound the treatment evaluation.
9. Having a life-threatening condition or immunocompromised (e.g., autoimmune deficiency syndrome, cancer, unstable angina, or myocardial infarction) within the last 6 months.
10. Unable to communicate or cooperate with the investigator due to language barriers, poor mental development, or impaired cerebral function.
11. Current participation in a clinical drug research study or recent participation in a clinical trial within 30 days of Baseline.
12. Using the following medications prior to Baseline:

    1. Antipruritics, including antihistamines within 3 days (72 hours).
    2. Topical corticosteroids, antibiotics or antifungal therapies within 4 weeks.
    3. Systemic corticosteroids, antibiotics or antifungal therapies within 12 weeks.
    4. Oral terbinafine or itraconazole within 12 weeks.
    5. Immunosuppressive medication or radiation therapy within 12 weeks.
    6. Any other topical medicated topical treatments to the treatment area(s) within 7 days.

       -

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2016-09; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Complete cure at Day 29 | Day 29
  The primary efficacy comparison between S2G6T-1 vs. rest of study arms will be based on the percentage of subjects at day 29 with complete cure of interdigital tinea pedis.mycological cure (i.e. negative dermatophyte culture and negative KOH) and clinical cure (i.e. absence of erythema, scaling and pruritus {scores of 0, each})
Reduction in Tinea pedis SymptomS through treatment period. | Day 8
  comparison of Patient Assessment between S2G6T-1 vs. rest of study arms will be based on the percentage of subjects at day 8 with achieving decrease from baseline in the total score for pruritus and burning.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen O Ashenfelter, MS, Study Chair — Cu-Tech, LLC
Locations (19):
- United States (19):
  - TCR Medical Corporation, San Diego, California
  - University Clinical Trials, Inc., San Diego, California
  - Tampa Bay Medical Research, Clearwater, Florida
  - Tory Sullivan, MD, PA, North Miami Beach, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - Mid Atlantic Research for Health, Baltimore, Maryland
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Skin Search of Rochester, Inc., Rochester, New York
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - DermResearch, Inc., Austin, Texas
  - J&S Studies, Inc, College Station, Texas
  - Suzanne Bruce & Associates, PA / The Center for Skin Research, Houston, Texas
  - Suzanne Bruce & Associates ,PA / The Center for Skin Research, Katy, Texas
  - DermResearch New Braunfels, New Braunfels, Texas
  - Endeavor Clinical Trials, PA, San Antonio, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah
  - The Education & Research Foundation Inc., Lynchburg, Virginia
  - Virginia Clinical Research Inc., Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Undecided